CLINICAL TRIAL: NCT00394602
Title: Chemoradiation-Induced Nausea and Emesis: A Prospective Study to Assess Patient Preferences and Quality of Life
Brief Title: Chemoradiation-Induced Nausea and Emesis: Quality of Life
Status: Terminated | Type: Observational
Why Stopped: Requested by PI during yearly Continuing Review
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2003-0529
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Gastric Cancer; Pancreatic Cancer; Cervical Cancer; Vulvar Cancer; Endometrial Cancer; Anal Cancer
Keywords: Gastric Cancer; Pancreatic Cancer; Cervical Cancer; Vulvar Cancer; Endometrial Cancer; Anal Cancer; Quality of Life; Questionnaire; Interview; Emesis; Nausea; Survey
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Endometrial Neoplasms; Anus Neoplasms; Vomiting; Nausea | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients receiving chemoradiation for abdominal-pelvic tumors.
  Interventions: Behavioral: Interview; Other: Questionnaire
- Caregiver Controls: Healthy controls with no prior cancer diagnosis.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Interview regarding perceptions of side effects that are related to chemoradiation treatment.
Other: Questionnaire — 3 Questionnaires regarding quality of life given during and after treatment, each taking about 20 minutes to complete.
  Other Names: Survey
  Groups: Patients

SUMMARY:
The primary objectives of this study are:

1. To assess the preferences of cancer patients scheduled to receive chemoradiation and caregiver controls for side-effects of chemoradiation.

   1. To compare preferences of cancer patients to those of healthy individuals.
   2. To compare how patients' preferences for side-effects of chemoradiation change over time.
2. To longitudinally assess the quality of life of cancer patients scheduled to receive chemoradiation.
3. To determine the impact of nausea and vomiting associated with chemoradiation on patients' quality of life and evaluate potential change throughout the duration of chemoradiation treatment.

DETAILED DESCRIPTION:
You will be interviewed about your perceptions of side effects that are related to your chemoradiation treatment. The interview will take about 20 minutes. You will be interviewed at the beginning of your chemoradiation treatment, 3 weeks after treatment starts, and at the first follow-up appointment after chemoradiation treatment ends.

Chemoradiation is a type of cancer treatment that involves both chemotherapy and radiation therapy.

You will also receive a packet of 3 questionnaires to complete at different times during and after treatment. The questionnaires include a quality of life survey that asks about physical, social, and emotional well-being, a self-report symptom evaluation that will ask whether you are experiencing any particular side effects and if so how much it bothers you, and a brief survey to asks questions about anxiety and distress.

The questionnaires should take about 20 minutes each to complete. The questionnaire packet will be given to patients at the beginning of chemoradiation treatment, 3 weeks after treatment starts, the last day of treatment, and at the first follow-up appointment after chemoradiation treatment ends. If the you do not have time to complete the questionnaires, a stamped, addressed envelop will be given so that you can mail the completed packet back to the research team.

Your participation in this research study will be over about 4-6 weeks after chemoradiation treatment ends.

This is an investigational study. Up to 208 individuals (104 patients and 104 caregivers) will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving 5 to 6-week course of chemoradiation for abdominal-pelvic tumors (gastric cancers, gastro-esophageal (GE) junction, pancreatic, cervix, vulvar, endometrial, or anal) using conventional fractionation [(180cGy-200cGy per day)]
2. Patients receiving concurrent abdominal-pelvic radiation and single agent or combination of cisplatin, paclitaxel, CPT-11, oxaliplatin or 5-FU, capecitabine, gemcitabine, or bevacizumab (Avastin).
3. Patients must be least 18 years of age
4. Controls must be individuals with no prior cancer diagnosis
5. Controls must be at least 18 years of age
6. Controls must be the caregivers of patients on this study

Exclusion Criteria:

1. Patients who do not have a diagnosis of cervix, endometrial, vulvar or anal cancer
2. Patients who are not scheduled to receive chemoradiation treatment
3. Patients who are not at least 18 years of age
4. Controls - individuals who have a prior diagnosis of cancer (with the exception of non-melanoma skin cancer)
5. Controls - individuals who are not at least 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving chemoradiation for abdominal-pelvic tumors and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2004-04-07 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Longitudinal Quality of Life + Symptom Assessment Data | Survey(s) & Interview(s) at baseline (beginning of chemoradiation treatment), 3 weeks after treatment starts, the last day of treatment, and at the first follow-up appointment after chemoradiation treatment ends.
  Quality of life survey instruments scored according to EORTC QLQ-C30 scoring manual. Patients and controls compared with respect to preference data. The control group preference data collected at only 1 time point, but patient preference data from each time point will be compared to these control group preference data.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte C. Sun, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org